CLINICAL TRIAL: NCT05333367
Title: MORPHEE : Mechanisms of Cell Death Induced by Extracorporeal Photochemotherapy
Acronym: MORPHEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022/679
Record Dates: First submitted 2022-04-04; First posted 2022-04-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous T-Cell Lymphoma; Graft Vs Host Disease; Graft Rejection
Keywords: Cell death; Extracorporeal Photochemotherapy
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing extracorporeal photochemotherapy (Other)
  Interventions: Other: Samples collection

INTERVENTIONS:
Other: Samples collection — Sampling of 2 samples on the extracorporeal photochemotherapy circuit, before and after sensitization with 8-MOP and UVA irradiation (without additional puncture)

SUMMARY:
The objective of this study is to describe the type of cell death induced by extracorporeal photochemotherapy, depending on the cell type, using a panel of complementary analysis techniques.

DETAILED DESCRIPTION:
Extracorporeal photochemotherapy (ECP) is a cell therapy used for its immunomodulation and tolerance induction capabilities. Its main indications are the control of graft-versus-host (GVH) disease in hematopoietic cell allografts, treatment and control of rejection in solid organ transplantation and the treatment of cutaneous T-cell lymphoma. Data on the mechanisms of action of ECP remains very patchy. This lack of data limits the discussion on therapeutic regimens by disease.

ECP consists of repeated apheresis sessions to collect leukocytes from the patient. The cells are then photosensitized, irradiated with UVA and reinjected into the patient in a closed circuit. In the context of GVH, induced cell death would stimulate the expansion of regulatory cells (Treg), restore a Th1/Th2 balance and decrease Th17 polarization. The ECP also allows the expansion of Treg in solid organ transplantation. Conversely, ECP would restore or activate an antitumor immune response in cutaneous T lymphoma.

The type of cells collected and treated would play a major role in the effects obtained. However, these hypotheses must be consolidated, in particular by detailing the initial role of cell death. Several questions remain, on the chronology of cell death in the different treated subpopulations, on the uptake by phagocytes, but especially on the type of cell death induced according to the cell type (necroptosis, apoptosis, pyroptosis, autophagy). The data generated will allow for validation or detail of the mechanisms of resolution of the inflammation and/or the anti-tumour effect observed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Treated with ECP for at least 1 month, for control of GVHD in hematopoietic cell allograft (acute or chronic GVHD), treatment and control of cellular or humoral rejection in solid organ transplantation (heart, lung, kidney) or in the treatment of cutaneous T-cell lymphoma

Exclusion Criteria:

* Subjects with limited legal capacity.
* Subjects judged by the investigator to be unlikely to comply with study procedures
* Subjects with no social security coverage.
* Pregnant women.
* Subjects still in the exclusion period of another study, or according to the national registry of clinical trial participants.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Type of cell death induced by 8-MOP sensitization and UVA irradiation | 24 hours
  Caspase-3 activation in Western blot
Type of cell death induced by 8-MOP sensitization and UVA irradiation | 24 hours
  Gasdermin D cleavage in Western blot
Type of cell death induced by 8-MOP sensitization and UVA irradiation | 24 hours
  MLKL (mixed lineage kinase domain-like pseudokinase) phosphorylation in Western blot

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No